CLINICAL TRIAL: NCT00984087
Title: rTMS for Adolescent and Young Adult Depression
Brief Title: rTMS for Adolescents and Young Adults
Acronym: JHU
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with recruitment and therefore funding has been pulled.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Irving Reti, Associate Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21284; NA_00021284 (Other: Johns Hopkins Institutional Review Board)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; TMS; adolescent; transcranial magnetic stimulation; MDD; Major depression; mood disorders
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mood Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active rTMS treatment (Experimental)
  Interventions: Device: TMS with Neurostar TMS Therapy System

INTERVENTIONS:
Device: TMS with Neurostar TMS Therapy System — 20 sessions with 1680 pulses per session at 10 Hz with a 4-second pulse train, stimulation at 100% motor threshold,
  Other Names: Neuronetics

SUMMARY:
rTMS is a promising, though largely untested, option for treating adolescent and young adult depression. This study hypothesizes that rTMS will safely and significantly alleviate depression and decrease suicidal ideation in adolescents and young adults based on previous studies.

DETAILED DESCRIPTION:
After signing consent and undergoing a thorough screening, participants will be administered rTMS 5 days per week for 4 consecutive weeks (a total of 20 sessions) as an add-on to their current antidepressant regime. Adolescents must be accompanied by a parent or legal guardian. We will monitor for depression, anxiety and suicidal ideation over the 4 weeks as well as 1 week following the last rTMS administration using rating scales. These scales will be given once a week, on Fridays, and will require roughly 40 minutes to complete. TMS sessions will last approximately 25 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MDD by a child and adolescent psychiatrist based on the DSM-IV, have a CDRS score of at least 60 or an HDRS score of at least 22 and have been suffering with depression during the current episode for at least 3 months
* Currently seeing a Johns Hopkins psychiatrist
* Excellent documentation of treatment resistance:

  * to at least 2 different antidepressant treatments, defined as resistance to a minimum of two antidepressant drug trials of adequate dose and duration in the current episode or previous episodes, adequacy being defined as a minimum level of three on the ATHF per antidepressant drug trial (those who have not completed antidepressant trials of adequate dose and duration due to intolerance to therapy may be included if they have demonstrated intolerance to three or more antidepressant medications in the current or a previous episode)
  * to at least one course of psychotherapy which did not result in significant alleviation of depressive symptoms
* No changes in medication dose or psychotherapy frequency over the previous 1 month
* Negative answers on the safety screening questionnaire for rTMS

Exclusion Criteria:

* History of substance abuse or dependence within the past six months (excluding nicotine and caffeine) or marked conduct disordered or oppositional behavior
* Any current unstable medical or surgical illness
* Bipolar Disorder
* Psychotic symptoms
* History of head injury or seizure or history of seizure in a first degree relative.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps
* History of frequent or severe headaches or migraines
* History of hearing loss or known history of cochlear implants.
* Pregnancy or not using a reliable method of birth control.
* Participation in another clinical trial within 30 days of this study
* Inability to locate and quantify a motor threshold (MT) as defined by the rTMS protocol
* Current use of drugs known to lower seizure threshold, such as stimulants, wellbutrin, bupropion, and certain tricyclics (e.g. clomipramine and maprotiline)
* Left-handed

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in depressive level after 4 weeks of rTMS compared with baseline scores. The Hamilton Depression Rating Scale (HDRS) will be used to measure changes in adolescents and young adults. | 4 weeks

SECONDARY OUTCOMES:
Change in depressive level using the CDRS (if adolescent) and HDRS (if young adult) at 1-week follow-up compared with baseline scores. | 5 weeks
Rates of remission (CDRS≤20; HDRS ≤10) and response (≥40% reduction in CDRS; ≥50% reduction in HDRS) at end of treatment and at follow-up. | 5 weeks
Measure across the 4 weeks of rTMS and at 1-week follow-up and compare with baseline scores the following: depressive symptoms, suicidal ideation, anxiety, and Clinical Global Impression-Severity Score (CGI-S). | 5 weeks
Safety of rTMS, as defined by maintained participant baseline pretreatment physical and neurological status. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Irving Reti, M.B.B.S, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States